CLINICAL TRIAL: NCT04985136
Title: A Randomized, Open-Label, Controlled, International Multi-Center Phase III Clinical Study of Camrelizumab Combined With Rivoceranib (Apatinib) Mesylate Versus Investigator's Choice of Regimen in Treatment of Patients With Hepatocellular Carcinoma (HCC) Who Have Been Treated With Immune Checkpoint Inhibitors (ICIs)
Brief Title: A Study of Camrelizumab Combined With Rivoceranib Mesylate Versus Investigator's Choice of Regimen in Treatment of Patients With Advanced Hepatocellular Carcinoma (HCC)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Sponsor R & D Strategy Adjustment
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-1210-III-330
Record Dates: First submitted 2021-07-15; First posted 2021-08-02 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2021-07

CONDITIONS: Advanced Hepatocellular Carcinoma (HCC)
MeSH Terms: interventions — apatinib; Sorafenib; regorafenib

STUDY DESIGN:
Intervention Model Description: Randomized，Open，Controlled, International Multi-Center
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- camrelizumab + Rivoceranib (Experimental)
  Interventions: Drug: camrelizumab；Rivoceranib
- Rivoceranib (Active Comparator)
  Interventions: Drug: Rivoceranib
- Sorafenib (Active Comparator)
  Interventions: Drug: Sorafenib
- Regorafenib (Active Comparator)
  Interventions: Drug: Regorafenib

INTERVENTIONS:
Drug: camrelizumab；Rivoceranib — Camrelizumab at 200 mg via intravenous administration (IV), once every 2 weeks (Q2W), in combination with 250 mg of rivoceranib mesylate, oral administration, once a day (QD)
  Arms: camrelizumab + Rivoceranib
Drug: Rivoceranib — Rivoceranib mesylate (750 mg, QD, po)
  Arms: Rivoceranib
Drug: Sorafenib — Sorafenib tosylate (400 mg, twice a day (BID), po)
  Arms: Sorafenib
Drug: Regorafenib — Regorafenib (160 mg, administer for 21 days then stop for 7 days, po)
  Arms: Regorafenib

SUMMARY:
This is a randomized, open-label, international, multi-center, phase III trial to evaluate the efficacy and safety of Camrelizumab Combined with Rivoceranib Mesylate versus Investigator's Choice of Regimen in Treatment of Patients with Hepatocellular Carcinoma (HCC)

ELIGIBILITY:
Inclusion Criteria:

1. Subject must participate voluntarily and sign the informed consent form;
2. Aged ≥ 18 years old, male or female;
3. Histopathologically confirmed hepatocellular carcinoma;
4. Has PD on treatment with prior anti-PD-1/PD-L1/CTLA-4 monoclonal antibody (mAb) administered either as monotherapy or as combination therapy.
5. No more than 2 lines of previous system treatment;
6. Be able to provide fresh or archived tumor tissue samples;
7. Patient with at least one measurable lesion (for Stage I);
8. Barcelona clinic liver cancer: Stage B or C;
9. Child-Pugh score: ≤ 7;
10. ECOG PS score of 0-1;
11. Life expectancy of ≥ 12 weeks;
12. Adequate organ function
13. Must take one medically approved contraceptive measure

Exclusion Criteria:

1. Patients with any active, known or suspected autoimmune disorder;
2. Patients who have used corticosteroids or other immunosuppressive agents for systemic treatment within 1 month prior to randomization;
3. With known severe allergic reactions to any other monoclonal antibodies;
4. Received previous camrelizumab or rivoceranib mesylate treatment;
5. Patients who discontinued ICIs treatment due to immune-related toxicity;
6. Patients with known CNS metastasis or hepatic encephalopathy;
7. Patients with liver tumor burden greater than 50% of total liver in volume, or patients who have previously undergone liver transplantation;;
8. Patients with symptomatic ascites or pleural effusion requiring paracentesis and drainage, or patients who have undergone ascites or pleural effusion drainage within 2 weeks before randomization;
9. Patients with other malignancies currently or within the past 5 years;
10. Patients with hypertension which cannot be well controlled by antihypertensives; history of hypertensive crisis or hypertensive encephalopathy;
11. Uncontrolled cardiac diseases or symptoms；
12. Known hereditary or acquired bleeding disorders;
13. Clinically significant bleeding symptoms or clear bleeding tendency;
14. Patients with gastrointestinal perforation or gastrointestinal fistula;
15. Patients with significant vascular invasions with a high possibility of fatal bleeding;
16. Patients with important arterial/venous thrombosis;
17. Patients experiencing toxicity caused by previous anti-tumor therapy that has not recovered to Grade ≤ 1;
18. Patients with active infection;
19. Patients with congenital or acquired immune deficiency;
20. Patients who received live vaccines within 28 days prior to randomization, or are expect to be vaccinated during the treatment period;
21. Patients with other potential factors that may affect the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2021-09-26 (Actual); Primary Completion 2021-12-29 (Actual); Study Completion 2021-12-29 (Actual)

PRIMARY OUTCOMES:
Stage I：Objective Response Rate（ORR） | 2.5 years
Stage II：Overall survival （OS） | 2.5 years

SECONDARY OUTCOMES:
Stage I：Overall survival （OS） | 2.5 years
Adverse Events（AEs） | 2.5 years
Stage II：Objective Response Rate（ORR） | 2.5 years
Disease Control Rate（DCR） | 2.5 years
Duration of Response（DoR） | 2.5 years
Progression-Free-Survival （PFS） | 2.5 years
time to progression （TTP） | 2.5 years
Pharmacokinetics (PK) Ctrough of camrelizumab | 2.5 years
Pharmacokinetics (PK) Ctrough of Apatinib | 2.5 years
Proportion of anti- camrelizumab antibody (ADA) | 2.5 years
Proportion of neutralizing antibody (Nab) | 2.5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China